CLINICAL TRIAL: NCT06939647
Title: Treprostinil Palmitil Inhalation Powder (TPIP) in Patients With Pulmonary Arterial Hypertension or Pulmonary Hypertension Associated With Interstitial Lung Disease
Brief Title: An Expanded Access Study to Assess Treprostinil Palmitil Inhalation Powder (TPIP) for Participants With Pulmonary Arterial Hypertension (PAH) and Pulmonary Hypertension Associated With Interstitial Lung Disease (PH-ILD)
Status: Available | Type: Expanded Access
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: TPIP EAP
Record Dates: First submitted 2025-04-11; First posted 2025-04-23 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Arterial Hypertension; Pulmonary Hypertension, Interstitial Lung Disease
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary; Lung Diseases, Interstitial

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Treprostinil Palmitil — Treprostinil Palmitil Inhalation Powder

SUMMARY:
The purpose of this study is to provide continued access to TPIP for participants who have successfully completed the open-label extension (OLE) studies of INS1009-203 for PAH or INS1009-212 for PH-ILD.

DETAILED DESCRIPTION:
Participants will receive TPIP 80 micrograms (μg), 160 μg, or 320 μg, inhalation single-dose capsules, orally, once daily (QD).

ELIGIBILITY:
Inclusion Criteria

* The participant is ineligible for or cannot be treated satisfactorily with alternative commercially available therapy for PAH or PH-ILD.
* Participant provides their informed consent to participate as per local requirements.
* Participant must have successfully completed the OLE INS1009-203 or INS1009-212 studies.
* Based on the treating physician's judgement on participant's medical history and an evaluation of the overall risk-benefit profile, the participant will be determined to be suitable for continued TPIP treatment within this program.
* Requests for the post-OLE INS1009-203 and INS1009-212 TPIP studies must originate from the investigators of INS1009-203 and INS1009-212 TPIP studies, respectively.
* Female participants must be postmenopausal (defined as no menses for 12 months without an alternative medical cause), surgically sterile, or using highly effective contraception (failure rate <1% per year when used consistently and correctly) from Day 1 to at least 90 days after the last dose.
* Male participants with female partners must adhere to contraception requirements to avoid potential exposure to the embryo/fetus based on the partner's reproductive status. For partners of childbearing potential, effective contraception must be used from Day 1 to at least 90 days after the last dose.

Exclusion Criteria:

• No specific exclusion criteria.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult